CLINICAL TRIAL: NCT06597773
Title: Online Patient Navigation Program for Timely Access to Supportive Care Services Among Patients With Breast Cancer
Brief Title: Online Patient Navigation Program for Patients With Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not possible to develop and implement the intervention due to lack of funding.
Sponsor: Medicos e Investigadores en la Lucha contra el Cancer de Mama (Other)
Responsible Party: Principal Investigator, Fernanda Mesa-Chavez, Principal Investigator, Medicos e Investigadores en la Lucha contra el Cancer de Mama
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECA-Navegacion
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Supportive Care in Cancer; Patient Navigation
Keywords: breast cancer; supportive care; patient navigation; online patient navigation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the intervention, the study will be open and participants will know which group they were randomized to. However, the study will be blinded to the statistician in order to reduce the risk of introducing bias when interpreting the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online patient navigation and supportive care referrals (Experimental): The intervention group will participate in an online patient navigation program designed to identify patients' nutrition, psychology, and sexology counseling needs, and to facilitate referrals and web-based systematic interventions to address these supportive care needs.
  Participants in this group will complete the study surveys at baseline (T1) and 4 weeks (T2) of follow-up.
  Interventions: Other: Online patient navigation and supportive care referrals
- In-person patient navigation and supportive care referrals (Active Comparator): The control group will participate in an in-person patient navigation program designed to identify patients' nutrition, psychology, and sexology counseling needs, and to facilitate referrals to in-person supportive care services.
  Participants in this group will complete the study surveys at baseline (T1) and 4 weeks (T2) of follow-up.
  Interventions: Other: In-person patient navigation and supportive care referrals

INTERVENTIONS:
Other: Online patient navigation and supportive care referrals — In the online patient navigation program, a navigator will use validated instruments to identify participants' need for nutrition, psychology, and sexology counseling, and will refer them to the required services. Referrals will be made to web-based, systematic supportive care resources consisting of pre-recorded videos led by specialists and which will be available on a study-specific website, allowing each participant to access the resources as soon as they receive a referral. Additionally, online support groups will be held monthly to complement the supportive care programs.
  Arms: Online patient navigation and supportive care referrals
Other: In-person patient navigation and supportive care referrals — In the in-person patient navigation program, a navigator will use validated instruments to identify participants' need for nutrition, psychology, and sexology counseling, and will refer them to the required services. Referrals will be made to supportive care services available at their healthcare institution.
  Arms: In-person patient navigation and supportive care referrals

SUMMARY:
The goal of this prospective 1:1 randomized controlled trial is to evaluate if an online patient navigation program, designed to identify targeted supportive care needs and to facilitate referrals and web-based interventions to address these needs, can increase patients' access to supportive care services, compared to traditional in-person patient navigation providing referrals to in-person supportive care services.

The main questions it aims to answer are:

* Does online patient navigation increase access to supportive care services among patients with breast cancer?
* Which are the barriers that hinder patients' access to the supportive care services they require?
* What is patients' level of satisfaction with online patient navigation?

Participants will:

* Participate in an online or in-person patient navigation program for 4 weeks
* Answer the study surveys at baseline and 4 weeks of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age ≥18 years
* Diagnosis of non-metastatic breast cancer
* Internet access at home or in their mobile phone
* Availability to answer the study surveys
* Provision of signed informed consent

Exclusion Criteria:

* Disease recurrence
* Inability to read or write

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09-21 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Access to supportive care services | 4 weeks
  Participants' rate of attendance to each of the supportive care services in study will be evaluated through a survey at 4 weeks of follow-up, which will assess each group's access to the recommended services, barriers encountered, and satisfaction with the navigation program.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Zambrano Hellion, San Pedro Garza García, Nuevo León, Mexico